CLINICAL TRIAL: NCT05611164
Title: SiD, an Assistant for Sperm Selection During Intracytoplasmic Sperm Injection in Medically Assisted Reproduction: Effect on Fertilization, Blastocyst Formation, Early Pregnancy Loss, and Consistent Practice. A Prospective Pilot Study.
Brief Title: Evaluation of SiD's System for Improving Assisted Reproduction Treatments
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IVF 2.0 Limited (Other)
Collaborators: New Hope Fertility Center Mexico (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P002-SP002
Record Dates: First submitted 2022-11-03; First posted 2022-11-09 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility | interventions — Sperm Injections, Intracytoplasmic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sperm selected by embryologist without software assistance (No Intervention): For each patient, oocytes collected following one ovarian stimulation cycle are randomly distributed in two groups ("no intervention" and "experimental" arms), in a sibling oocyte study design. In the "no intervention" arm, the individual spermatozoa for injection are selected subjectively by the embryologist.
- Sperm selected with AI assistant SiD (Experimental): For each patient, oocytes collected following one ovarian stimulation cycle are randomly distributed in two groups ("no intervention" and "experimental" arms), in a sibling oocyte study design. In the "experimental" arm, the spermatozoa selection for injection is performed based on the recommendation of the AI assistant SiD.
  Interventions: Device: Software assisted selection of individual spermatozoa for intracytoplasmic sperm injection

INTERVENTIONS:
Device: Software assisted selection of individual spermatozoa for intracytoplasmic sperm injection — Half of the oocytes will be injected with a sperm selected with SiD's assistance
  Arms: Sperm selected with AI assistant SiD

SUMMARY:
According to the WHO, infertility affects 15% of reproductive age couples worldwide. Among the assisted reproductive technologies available for patients with infertility, intracytoplasmic sperm injection (ICSI) has become one of the most widely employed and is now thought to be the most common method for oocyte insemination outside of the human body.

ICSI entails the selection of an individual sperm cell and its injection directly into an oocyte. Usually, an embryologist performs the selection of the individual sperm cell to inject by subjectively observing the morphology and progression of the candidate spermatozoon. Subjectivity and time constrains, however, suggest the best possible candidate might not always be selected. Further optimization of ICSI technology remains a significant goal, yet the majority of approaches proposed in the literature have returned mixed results. The deployment of an artificial intelligence (AI) software capable of detecting and non-invasively predicting the value of individual spermatozoa in real time could significantly improve ICSI.

SiD (IVF 2.0 Ltd, London, UK) is a software designed to identify, evaluate, and assist in the spermatozoon selection process ahead of ICSI. SID uses a mathematical model to evaluate individual spermatozoa in real-time according to their motility patterns (for instance velocity, linearity, straightness) and their morphology. The software has been developed by making use of retrospective data analysis, but its prospective evaluation is still pending.

With the above in mind, this study intends to address the following question: can the use of a software assistant for the selection of individual sperm cells for injection (SiD), improve ICSI outcomes (oocyte fertilization, embryo development and quality, embryo ploidy, pregnancy, and live birth)? Patients with a clinical indication for undergoing ICSI will be prospectively enrolled into the study. Following ovarian stimulation, the oocytes retrieved from each patient will be randomly split into two groups and inseminated by ICSI using sperm selected either subjectively by an embryologist (control group) or by the software assistant SiD (experimental group). Embryos will be allowed to develop for up to six days and until blastocyst formation assessments are completed. Embryos might be subjected to cytogenetic screening or used for embryo transfer according to patient needs. The recorded outcomes will be anonymized prior to statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Participant's age between 18 and 40 years of age.
* Informed consent signed by the patient before treatment.
* IVF treatments with medical or embryology indication to perform ICSI.
* Cycles with at least 2 oocytes in Metaphase II.
* Fresh ejaculated motile sperm.
* Fresh oocytes.
* Selection of sperm using a 7% or 10% PVP solution.
* Presence of motile sperm at the time of sperm selection for ICSI.
* Videos recorded with a total magnification of 200x.

Exclusion Criteria:

* Patients diagnosed with recurrent pregnancy loss.
* Spermatozoa extracted by testicular biopsy.
* Frozen/thawed spermatozoa.
* Frozen/thawed oocytes in any case.
* That the recommendations for use of SiD have not been fully followed.
* Poor quality of saved ICSI video.
* Inability to reliably trace sperm-oocyte-embryo throughout the process.
* Oocytes that are not in Metaphase II.
* Patients with immotile sperm

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-09-05 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Fertilization rate | 16-18 hours after ICSI
  Rate of oocytes that present two pronuclei or cell division
Blastocyst formation rate | around 120 hours after ICSI
  Rate of oocytes that have a defined trophectoderm and inner cell mass
Usable blastocyst formation rate | around 120 hours after ICSI
  Rate of oocytes that have a blastocyst that is transferable accoring to its quality

SECONDARY OUTCOMES:
Ploidy status | trophectoderm biopsy is performed around 120 hours after ICSI
  euploid rate (when available)
Biochemical pregnancy | 2 weeks after blastocyst transference
  human beta chorionic gonadotropin
Clinical pregnancy | 6 weeks after blastocyst transference
  Presence of heartbeat

CONTACTS AND LOCATIONS:
Locations (2):
- Mexico (2):
  - New Hope Fertility Center, Guadalajara, Jalisco
  - New Hope Fertility Center, Mexico City

IPD SHARING:
Plan to Share IPD: No